CLINICAL TRIAL: NCT03645057
Title: ASPIRE: DETERIMINING THE IMPACT OF CRISABOROLE (Eucrisa) AND TACROLIMUS 0.03% ON PATIENT-REPORTED OUTCOMES AND CAREGIVER BURDEN IN CHILDREN WITH ATOPIC DERMATITIS
Brief Title: ASPIRE: PROs & Caregiver Burden in Children With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Julie Ryan Wolf, Associate Professor of Dermatology & Radiation Oncology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRB73062
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole; Tacrolimus; Ointments

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, cross-sectional study to monitor the effects of crisaborole and tacrolimus 0.03% on patient-reported outcomes and caregiver burden in children (ages 2 to 15 years, inclusive) with ≤ moderate atopic dermatitis over a 12 week period of time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Crisaborole (Experimental): The topical treatment will be applied to all affected areas twice daily for 12 weeks.
  Interventions: Drug: Crisaborole
- Tacrolimus 0.03% (Active Comparator): The topical treatment will be applied to all affected areas twice daily for 12 weeks.
  Interventions: Drug: Tacrolimus 0.03% Ointment

INTERVENTIONS:
Drug: Crisaborole — This topical ointment is FDA-approved to treat atopic dermatitis of moderate or less severity in children. Subjects will apply the topical ointment to all affected areas twice daily for 12 weeks.
  Other Names: Eucrisa
  Arms: Crisaborole
Drug: Tacrolimus 0.03% Ointment — This topical ointment is FDA-approved to treat atopic dermatitis in children. Subjects will apply the topical ointment to all affected areas twice daily for 12 weeks.
  Other Names: Protopic
  Arms: Tacrolimus 0.03%

SUMMARY:
This is an open-label, randomized, cross-sectional study to monitor the effects of crisaborole and tacrolimus 0.03% on patient-reported outcomes and caregiver burden in children (ages 2 to 15 years, inclusive) with ≤ moderate atopic dermatitis over a 12 week period of time. The goal of this study is to detect changes in PROs and caregiver burden during treatment for atopic dermatitis of moderate or less severity. The study design will allow us to correlate PROs and caregiver burden with treatment response and disease improvement in children.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a common, chronic skin disease affecting 20% of children and 10% of adults worldwide (1-3). Children with AD often develop the disease within the first five years of life, which is a critical time for physical and psychosocial development (4). AD impacts an individual's physical, mental, and social health. Anxiety, itch, sleep disturbance, and depression have been associated with low quality of life scores. Childhood AD also affects the emotional, financial, physical, and social well-being of parents or caregivers (4). Individuals caring for a child with AD report sleep deprivation, poor social support, and stress about parenting (1, 4). Utilizing patient-reported outcomes (PROs) in clinic can provide meaningful data to monitor disease activity and response to different interventions, with the ultimate goal to improve quality of life for the patient and their family members or caregivers. Additionally, PROs can help us better understand the burden of AD. It is still unclear which PROs are most relevant for atopic dermatitis. This study will evaluate the utility of several PROs to monitor response to two different topical ointments, crisaborole (Eucrisa™) and tacrolimus 0.03%, to better understand the impact of these two non-steroidal topical treatments on overall health of children with AD of moderate or less severity and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

Pediatric Subjects:

1. Male and female subjects of inclusive ages of 2 to 15 years (inclusive) at screening visit.
2. Diagnosis of ≤moderate atopic dermatitis or eczema (ISGA 2 or 3 and ≥3% BSA, excluding scalp).
3. If subject is taking or prescribed antihistamines, subject must be on stable dose of antihistamines.
4. If subject is taking or prescribed topical steroids, subject must be on stable dose of topical steroids.
5. If taking a systemic anti-inflammatory medication for atopic dermatitis or other condition, subject must be on stable dose of the systemic anti-inflammatory medication for six weeks prior to enrollment.
6. If subject is currently taking or prescribed tacrolimus or crisaborole, or other steroid-sparring medication, subject must agree to two week (i.e., 14 days) washout period prior to randomization and Baseline Assessment for study.
7. Caregiver (i.e., adult parent or guardian) must agree to participate in the study with the patient.

e) Subject must be able to read and speak English. f) Subject ages ≥8 years, is able to give assent.

Caregiver Subjects:

1. Subject must be at least 18 years old and the parent or guardian of the eligible pediatric subject.
2. Subject must be able to read and speak English.
3. Subject must be able to give informed consent.

Exclusion Criteria:

1. Pediatric subjects <2 years old or >15 years old are not eligible for participation in this study.
2. Pediatric subjects with a diagnosis with another skin disease (i.e., not atopic dermatitis or eczema) are excluded to prevent confounding of results.
3. Pediatric subjects currently on systemic anti-inflammatory therapy for atopic dermatitis or other indication are excluded.
4. Caregiver subject <18 years old are excluded.
5. Pediatric subject participation without caregiver participation is not allowed.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie R Wolf, PhD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Dermatology, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled child patients and caregiver (i.e., parent) dyads. Child patients with mild to moderate atopic dermatitis were enrolled based on the inclusion and exclusion criteria (see eligibility criteria). A caregiver (i.e., parent) of each child had to agree to participate in the trial.
Pre-assignment Details: There were 47 patient/caregiver dyads (i.e., 94 subjects total = 47 child patients with 47 caregivers). If the child patient was already actively using cisaborole or tacrolimus 0.03% for their atopic dermatitis, child patient underwent a two week wash out before baseline assessment and randomization. One dyad was lost to follow up prior to randomization. Therefore, 46 dyads were randomized to one of the two study arms.
Groups:
- Crisaborole-children: The topical treatment will be applied to all affected areas twice daily for 12 weeks.
  Crisaborole: This topical ointment is FDA-approved to treat atopic dermatitis of moderate or less severity in children. Subjects will apply the topical ointment to all affected areas twice daily for 12 weeks. At each study visit, the child patient had their clinical severity of atopic dermatitis rated by a clinician and the child patients completed five outcome measures (PROMIS Pediatric Itch (Static Form), PROMIS Pain Interference (CAT), Children's Dermatology Life Quality Index, PROMIS Anxiety (CAT), PROMIS Depression (CAT).
- Tacrolimus-children: The topical treatment will be applied to all affected areas twice daily for 12 weeks.
  Tacrolimus 0.03% Ointment: This topical ointment is FDA-approved to treat atopic dermatitis in children. Subjects will apply the topical ointment to all affected areas twice daily for 12 weeks. At each study visit, the child patient had their clinical severity of atopic dermatitis rated by a clinician and the child patients completed five outcome measures (PROMIS Pediatric Itch (Static Form), PROMIS Pain Interference (CAT), Children's Dermatology Life Quality Index, PROMIS Anxiety (CAT), PROMIS Depression (CAT).
- Crisaborole-caregivers: This was a dyad study. A caregiver was enrolled for each child. The caregiver completed three outcome measures at each study visit (Children's Sleep Habits Questionnaire, Family Dermatology Life Quality Index (FDLQI), and Caregiver Burden Inventory).
- Tacrolimus-caregivers: This was a dyad study. A caregiver was enrolled for each child. The caregiver completed three outcome measures at each study visits (Children's Sleep Habits Questionnaire, Family Dermatology Life Quality Index (FDLQI) and Caregiver Burden Inventory).
Period: Randomization to Baseline
Arm/Group | Crisaborole-children | Tacrolimus-children | Crisaborole-caregivers | Tacrolimus-caregivers
Started (46 patient/caregiver dyads were randomized to crisaborole or tacrolimus 0.03% study arms (i.e., 92 subjects total = 46 child patients and 46 caregivers).) | 23 | 23 | 23 | 23
Completed (One dyad (i.e., 1 child patient with 1 caregiver) was lost to followup after randomization (i.e., crisaborole arm) but before baseline assessment. This dyad was one that required a washout prior to baseline assessment. The Baseline Assessment included clinician-rated severity of the child patient's atopic dermatitis. completion of five outcome measures by the child patient, and completion of three outcome measures by the caregiver.) | 22 | 23 | 22 | 23
Not Completed | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Period: Baseline to Six Weeks
Arm/Group | Crisaborole-children | Tacrolimus-children | Crisaborole-caregivers | Tacrolimus-caregivers
Started (45 dyads (i.e., 90 subjects total = 45 child patients and 45 caregivers) completed Baseline Assessment. Child patient used the assigned study medication for 6 weeks (baseline visit to 6 week study visit). The 6 week study visit included clinician-rated severity of child patient's atopic dermatitis, completion of five outcome measure by the child patient, and completion of three outcome measure by the caregiver.) | 22 | 23 | 22 | 23
Completed (Child subjects used their assigned topical medication for 6 weeks (baseline to 6 week study visits). 1 dyad (i.e., 2 subject total = 1 child patient and 1 caregiver) in the crisaborole arm withdrew from the study because the caregiver no longer wanted to participate. 5 dyads (i.e., 10 subject total = 5 child patients and 5 caregivers) in the crisaborole arm were lost to followup. 1 dyad (i.e., 2 subjects total = 1 child patient and 1 caregiver) in the tacrolimus arm was lost to follow-up.) | 16 | 21 | 16 | 21
Not Completed | 6 | 2 | 6 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 5 | 2 | 5 | 2
Period: 6 Weeks to 12 Weeks
Arm/Group | Crisaborole-children | Tacrolimus-children | Crisaborole-caregivers | Tacrolimus-caregivers
Started (37 dyads (i.e., 74 subject total = 37 child patients and 37 caregivers) completed the 6 week assessment. The child patients continued using their assigned topical medication for 6 weeks until the 12 week study visit.) | 16 | 21 | 16 | 21
Completed (36 dyads (i.e., 72 subjects total = 36 child patients and 36 caregivers) completed their assigned topical medication for 12 weeks and completed the 12 week study visit. 1 dyad (i.e., 2 subject total = 1 child patient and 1 caregiver) in the tacrolimus arm was lost to followup. The 12 week study visit included clinician-rated severity of the child patient's atopic dermatitis, completion of five outcome measures by the child patient, and completion of three outcome measures by the caregiver.) | 16 | 20 | 16 | 20
Not Completed | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Crisaborole-children: The topical treatment will be applied to all affected areas twice daily for 12 weeks.
  Crisaborole: This topical ointment is FDA-approved to treat atopic dermatitis of moderate or less severity in children. Subjects will apply the topical ointment to all affected areas twice daily for 12 weeks.
- Tacrolimus-children: The topical treatment will be applied to all affected areas twice daily for 12 weeks.
  Tacrolimus 0.03% Ointment: This topical ointment is FDA-approved to treat atopic dermatitis in children. Subjects will apply the topical ointment to all affected areas twice daily for 12 weeks.
- Crisaborole-caregiver; Tacrolimus-caregiver: This was a dyad study. A caregiver was enrolled for each child.
- Total: Total of all reporting groups
Arm/Group | Crisaborole-children | Tacrolimus-children | Crisaborole-caregiver | Tacrolimus-caregiver | Total
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The children and caregiver groups were analyzed separately.
  years
    children: number analyzed (Participants) | 23 | 23 | 0 | 0 | 46
    children | 9.3 (3.4) | 8.3 (4.1) |  |  | 8.8 (3.7)
    caregivers: number analyzed (Participants) | 0 | 0 | 23 | 23 | 46
    caregivers |  |  | 37.3 (5.9) | 36.9 (8.4) | 37.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 19 | 19 | 64
  Male | 8 | 12 | 4 | 4 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 5 | 2 | 13
  Not Hispanic or Latino | 18 | 21 | 17 | 21 | 77
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 9 | 9 | 36
  White | 6 | 10 | 8 | 11 | 35
  More than one race | 3 | 2 | 1 | 1 | 7
  Unknown or Not Reported | 4 | 1 | 4 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 23 | 23 | 92

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Children's PROMIS Pediatric Itch Short-Form
Description: This is a patient-reported outcome measure for Itch in pediatric patients that consists of 8 fixed items items, spanning four domains (general, activity, mood/sleep, and scratching behavior). Each item is scored on using 1 = No Itch, 2 = Mild, 3 = Moderate, 4 = Severe, and 5 = Very Severe. The range of the scale is 1 to 5 with higher numbers indicating worse outcome. A total score, representing overall itch-related quality of life, is scored by taking the average (i.e., divide by 8) of the sum of all 8 items. Therefore, total itch scores range between 1 and 5, with higher scores indicating worse impact of itch on quality of life. The measure was completed electronically on an iPad using REDCap.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Tacrolimus 0.03%
Number analyzed (Participants) | 16 | 20
score on a scale | -0.3 (0.8) | -0.4 (0.8)
Statistical Analysis 1: Comparison: Crisaborole vs Tacrolimus 0.03%; Test type: Superiority; p = 0.433, Wilcoxon rank sum test

2. Primary Outcome: Mean Change in PROMIS Pain Interference-Children (Adaptive Test)
Description: This is a patient reported outcome measure for pain interference in pediatric patients. This is a computer adaptive test consisting of 4-12 questions related to how pain interferes with daily activities. The number of questions a patient answers depends on how he or she answers each question. The overall domain score ranges from 0 to100 with a score of 50 representing the average score for the general population. Higher scores indicate greater pain interference. A score above 55 is considered "clinically significant" for each domain. A score change of 5 or more is considered a clinically important change in domain severity. This measure was completed electronically on an iPad using REDCap.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Crisaborole | Tacrolimus 0.03%
Number analyzed (Participants) | 16 | 20
T-score | -6.4 (10.4) | -6.8 (9.3)
Statistical Analysis 1: Comparison: Crisaborole vs Tacrolimus 0.03%; Test type: Superiority; p = 0.836, Wilcoxon rank sum test

3. Secondary Outcome: Mean Change in Children's Dermatology Life Quality Index
Description: This patient-reported outcome measure will be completed using an iPad. The 10-item questionnaire designed for use in parents of children (i.e., ages 4-17) to obtain information on children's quality of life. Each question relates to a component of quality of life: Symptoms/Feelings (items 1-2); Leisure (items 4-6); School (item 7); Relationships (items 3-8); Sleep (item 9), and Treatment (item 10). Children answer each question using a 4-point scale: Not at all = 0, A Little = 1, Quite A Lot = 2, Very Much = 3. The scores from each item are summed to create a severity burden score (i.e., minimum score = 0; maximum score = 30). Higher the scores, the greater burden on quality of life. The scores represent degree of severity burden on quality of life: No effect = 0-1; Small effect = 2-6; Moderate effect = 7-12; Very large effect = 13-18; and Extremely large effect = 19-30.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Tacrolimus 0.03%
Number analyzed (Participants) | 16 | 20
score on a scale | -1.1 (4.0) | -3.6 (4.2)
Statistical Analysis 1: Comparison: Crisaborole vs Tacrolimus 0.03%; Test type: Superiority; p = 0.073, Wilcoxon rank sum test

4. Secondary Outcome: Mean Change in Children's Sleep Habits Questionnaire
Description: This patient-reported outcome measure was completed by the caregiver using an iPad. This is a validated 22 item questionnaire consisting of 4 subscales: Bedtime, Sleep Behavior, Waking During the Night, and Morning Wake Up. The patient/parent will answer each item choosing from: "Always" if something occurs every night; "Usually" if it occurs 5 or 6 times a week; "Sometimes" if it occurs 2 to 4 times a week; "Rarely" if it occurs once a week; and "Never" if it occurs less than once a week. Each question is scored on a 3-point scale as 1 = Usually and Always (5-7 times/week); 2 = Sometimes" (2-4 times/week); or 3 = Rarely and Never (0-1 time/week). The scores are combined from each subscale to generate a Total Sleep Disturbance Score, which can range from 22 (minimum) to 66 (maximum). The higher the score, the greater the sleep disturbance. A Total Sleep Disturbances score over 28 represent clinically significant sleep disturbance.
Time Frame: Baseline to 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Tacrolimus 0.03%
Number analyzed (Participants) | 16 | 20
score on a scale | -1.7 (6.0) | -1.3 (7.0)
Statistical Analysis 1: Comparison: Crisaborole vs Tacrolimus 0.03%; Test type: Superiority; p = 0.989, Wilcoxon rank sum test

5. Secondary Outcome: Mean Change in PROMIS Anxiety-children (Adaptive Test)
Description: This patient-reported outcome measure will be completed by the child patient electronically on an iPad using computer adaptive test (CAT). The CAT consists of 4-12 questions on feelings related to anxiety. The number of questions a patient answers depends on how he or she answers each question. The domain score is a t-score ranging from 0 to 100 with a score of 50 representing the average score for the general population. Higher scores indicate greater anxiety. A score above 55 is considered "clinically significant" for each domain. A score change of 5 or more is considered a clinically important change in domain severity. This PRO was completed electronically on an iPad using REDCap.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Crisaborole | Tacrolimus 0.03%
Number analyzed (Participants) | 16 | 20
T-score | -5.0 (9.8) | -6.8 (8.4)
Statistical Analysis 1: Comparison: Crisaborole vs Tacrolimus 0.03%; Test type: Superiority; p = 0.565, Wilcoxon rank sum test

6. Secondary Outcome: Mean Change in PROMIS Depressive Symptoms-Pediatric (Adaptive Test)
Description: This patient-reported outcome measure s will be completed by the child patient electronically on an iPad using computer adaptive test (CAT). The CAT consists of 4-12 questions on feelings related to depressive symptoms. The number of questions a patient answers depends on how he or she answers each question. The domain score is a t-score ranging from 0 to 100 with a score of 50 representing the average score for the general population. Higher scores indicate greater depressive symptoms. A score above 55 is considered "clinically significant" for each domain. A score change of 5 or more is considered a clinically important change in domain severity. This PRO was completed electronically on an iPad using REDCap.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Crisaborole | Tacrolimus 0.03%
Number analyzed (Participants) | 16 | 20
T-score | -4.0 (7.4) | -5.8 (9.5)
Statistical Analysis 1: Comparison: Crisaborole vs Tacrolimus 0.03%; Test type: Superiority; p = 0.479, Wilcoxon rank sum test

7. Secondary Outcome: Mean Change in Children's Eczema Area & Severity Index (EASI)
Description: Clinician rated the severity of atopic dermatitis using the EASI. The EASI is a tool used to measure the extent (area) and severity of AD. It does not include a grade for dryness or scaling and includes only inflamed areas. The area score is a 7-point scale representing the percentage of skin affected by AD for each body region. The severity score is recorded for each of the four regions of the body and is the sum of the intensity scores for four signs. The four signs include redness, thickness, scratching, and lichenification. The intensity scores are performed using a 4-pont scale. The final EASI score is the sum of the total scores for each region. Add up the total scores for each region to determine the final EASI score. The minimum EASI score is 0 and the maximum EASI score is 72. Higher scores represent worse AD severity.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Tacrolimus 0.03%
Number analyzed (Participants) | 16 | 20
score on a scale | -2.4 (2.9) | -1.9 (3.0)
Statistical Analysis 1: Comparison: Crisaborole vs Tacrolimus 0.03%; Test type: Superiority; p = 0.577, Wilcoxon rank sum test

8. Other Pre Specified Outcome: Mean Change in Caregiver Burden Inventory
Description: The CBI is a 24-item, five-subscale Caregiver Burden Inventory (CBI) and demonstrates its use as a diagnostic tool for caregiver burden. The five subscales include: Time Dependency, Development, Physical Health, Emotional Health, and Social Relationships. Each subscale contains 4-5 items which are statements of feelings. Caregivers use a 5-point scale, anchored by "0" = "Never" and "4" = "Nearly Always", to show how often the statement describes his/her feelings. Overall scores can range from 0 (minimum) to 96 (maximum), where a score near or above 36 indicates significant burden. Higher scores indicate greater caregiver burden (i.e., worse outcome). All subscales have a maximum score of 20, except Physical Health which has a maximum score of 16. Subscale scores and item scores help identify the underlying cause of caregiver burden. This measure will be completed electronically on an iPad using REDCap.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Tacrolimus 0.03%
Number analyzed (Participants) | 16 | 20
score on a scale | -1.3 (7.2) | -4.2 (6.8)
Statistical Analysis 1: Comparison: Crisaborole vs Tacrolimus 0.03%; Test type: Superiority; p = 0.439, Wilcoxon (Mann-Whitney)

9. Other Pre Specified Outcome: Mean Change in Family Dermatology Life Quality Index
Description: The FDLQI is a 10-item questionnaire designed for adult family members of a patient with a skin disease. It measures the impact of the patient's skin disease on the family member's quality of life. The caregiver will answer each question using a 4-point scale: Not at all = 0, A Little = 1, Quite A Lot = 2, Very Much = 3. The scores from each item are summed to create a severity burden score (i.e., minimum score = 0; maximum score = 30). Higher scores indicate worse quality of life. The scores represent degree of severity burden on quality of life: No effect = 0-1; Small effect = 2-6; Moderate effect = 7-12; Very large effect = 13-18; and Extremely large effect = 19-30. This measure will be completed electronically on an iPad using REDCap.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole | Tacrolimus 0.03%
Number analyzed (Participants) | 16 | 20
score on a scale | -2.6 (4.0) | -3.6 (2.9)
Statistical Analysis 1: Comparison: Crisaborole vs Tacrolimus 0.03%; Test type: Superiority; p = 0.242, Wilcoxon rank sum test

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Adverse events were not collected for the caregivers.
Arm/Group | Crisaborole-children | Tacrolimus-children
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/21
Other Adverse Events (participants affected / at risk) | 2/16 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crisaborole-children (N=16) | Tacrolimus-children (N=21)
molluscum (Infections and infestations) | 0 | 1
lacerations and bruising (Injury, poisoning and procedural complications) | 0 | 1
nose bleed (Vascular disorders) | 1 | 0
atopic dermatitis flare (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT03645057/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03645057/ICF_001.pdf